CLINICAL TRIAL: NCT02789345
Title: An Open-Label, Multicenter, Phase 1 Study With Expansion Cohorts of Ramucirumab or Necitumumab in Combination With Osimertinib in Patients With Advanced T790M-Positive EGFR-Mutant Non-Small Cell Lung Cancer After Progression on First-Line EGFR TKI Therapy
Brief Title: A Study of Ramucirumab (LY3009806) or Necitumumab (LY3012211) Plus Osimertinib in Participants With Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16357; I4T-MC-JVDL (Other: Eli Lilly and Company); 2015-005296-25 (EudraCT Number)
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: T790M; epidermal growth factor receptor (EGFR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; necitumumab; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Ramucirumab + Osimertinib (Experimental): Dose Finding: Participants received Ramucirumab 10 milligrams/kilogram (mg/kg) given intravenously (IV) on day 1 every 2 weeks and osimertinib 80 milligrams (mg) given orally daily during each 14-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Osimertinib
- Arm B: Necitumumab + Osimertinib (Experimental): Dose Finding: Participants received Necitumumab 800 mg given IV on days 1 and 8 every 3 weeks and osimertinib 80 mg given orally daily during each 21 day cycle.
  Interventions: Drug: Necitumumab; Drug: Osimertinib
- Cohort A: Ramucirumab + Osimertinib (Experimental): Dose Expansion: Participants received Ramucirumab 10 mg/kg given IV on day 1 every 2 weeks and osimertinib 80 mg given orally daily during each 14-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Osimertinib

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: Arm A: Ramucirumab + Osimertinib; Cohort A: Ramucirumab + Osimertinib
Drug: Necitumumab — Administered IV
  Other Names: LY3012211
  Arms: Arm B: Necitumumab + Osimertinib
Drug: Osimertinib — Administered orally
  Other Names: AZD9291

SUMMARY:
The main purpose of this study is to evaluate the safety of ramucirumab or necitumumab in combination with osimertinib in participants with non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of NSCLC with at least 1 measurable lesion assessable using standard techniques by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
* Have T790M-positive status using a test validated and performed locally after disease progression on EGFR tyrosine kinase inhibitor (TKI) treatment.
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 at the time of enrollment.
* Have serum albumin that is ≥25 grams per liter at the time of enrollment.
* Have adequate organ function, with all screening labs performed within 7 days of treatment initiation.
* Have a life expectancy of ≥3 months.
* Have resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior systemic cancer therapy, surgery, or radiotherapy to Grade ≤1 by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

Exclusion Criteria:

* Previous treatment with an EGFR monoclonal antibody (except for past treatment for squamous cell carcinoma of head and neck or metastatic colorectal cancer).
* Previous treatment with osimertinib or third generation EGFR TKIs.
* Participants with symptomatic or growing brain metastases less than 4 weeks prior to enrollment.
* History of drug-induced interstitial lung disease (ILD), ILD, or radiation pneumonitis requiring treatment with steroid prior to study enrollment, or any evidence of clinically active ILD.
* Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment. Participants with a history of gross hemoptysis (defined as bright red blood of ≥1/2 teaspoon) within 2 months prior to enrollment are excluded.
* Have experienced any arterial thrombotic event or arterial thromboembolic event, including myocardial infarction, unstable angina (history or evidence of current clinically relevant coronary artery disease of current ≥Class III as defined by Canadian Cardiovascular Society Angina Grading Scale or congestive heart failure of current ≥Class III as defined by the New York Heart Association), cerebrovascular accident, or transient ischemic attack, within 6 months prior to enrollment.
* Have a history of deep vein thrombosis, pulmonary embolism, or any other significant venous thromboembolism (venous catheter thrombosis or superficial venous thrombosis not considered "significant") during the 3 months prior to study enrollment. Participants with venous thromboembolism occurring 3 to 6 months prior to study enrollment are allowed, if being treated with low molecular weight heparin.
* Have a history of gastrointestinal perforation and/or fistula within 6 months prior to enrollment.
* Have a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Have uncontrolled hypertension, as defined in CTCAE Version 4.0, prior to initiating study treatment, despite antihypertensive intervention. CTCAE Version 4.0 defines uncontrolled hypertension as Grade >2 hypertension; clinically, the participant continues to experience elevated blood pressure (systolic >160 millimeters of mercury [mmHg] and/or diastolic >100 mmHg) despite medications.
* Are receiving chronic therapy with any of the following medications within 7 days prior to enrollment:

  * nonsteroidal anti-inflammatory agents (NSAIDs; such as indomethacin, ibuprofen, naproxen, or similar agents).
  * other anti-platelet agents (such as clopidogrel, ticlopidine, dipyridamole, or anagrelide).
* Have radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Have radiographic evidence of pulmonary intratumor cavitation, regardless of tumor histology.
* Are receiving concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, chemoembolization, or targeted therapy or radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks prior to enrollment.
* Have abnormal cardiac findings.
* Have undergone chest irradiation within 2 weeks prior to study drug administration, have not recovered from all radiation-related toxicities, or requires corticosteroids. A 2-week washout is permitted for focal palliative radiation to non-central nervous system disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif, France
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheong Ju-City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- [Derived] Yu HA, Paz-Ares LG, Yang JC, Lee KH, Garrido P, Park K, Kim JH, Lee DH, Mao H, Wijayawardana SR, Gao L, Hozak RR, Chao BH, Planchard D. Phase I Study of the Efficacy and Safety of Ramucirumab in Combination with Osimertinib in Advanced T790M-positive EGFR-mutant Non-small Cell Lung Cancer. Clin Cancer Res. 2021 Feb 15;27(4):992-1002. doi: 10.1158/1078-0432.CCR-20-1690. Epub 2020 Oct 12. PMID 33046516
- See also: A Study of Ramucirumab (LY3009806) or Necitumumab (LY3012211) Plus Osimertinib in Participants With Lung Cancer — https://trials.lillytrialguide.com/en-US/trial/4jipcrdi0g6CmmMMe8mUyI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of the dose-finding portion (Phase 1a) and the dose-expansion portion (Phase 1b)
  * Phase 1a, Arm A = combination of ramucirumab and osimertinib; Arm B = combination of necitumumab and osimertinib
  * Phase 1b included one cohort, the expansion of Arm A with additional participants enrolled i.e., Cohort A, a combination of ramucirumab and osimertinib. Per Protocol, all outcomes for a combination of ramucirumab and osimertinib were analyzed under a single arm i.e., Arm A/Cohort A
Pre-assignment Details: Participants who did not "complete" study were those who discontinued study treatment by the time of study completion.
Groups:
- Arm A: Ramucirumab + Osimertinib; Cohort A: Ramucirumab + Osimertinib: Participants received Ramucirumab 10 mg/kg given IV on Day 1 every 2 weeks and osimertinib 80 mg given orally daily during each 14-day cycle. All participants were treated until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Arm B: Necitumumab + Osimertinib: Participants received Necitumumab 800 mg given IV on Days 1 and 8 every 3 weeks and osimertinib 80 mg given orally daily during each 21-day cycle. All participants were treated until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
Period: Overall Study
Arm/Group | Arm A: Ramucirumab + Osimertinib | Arm B: Necitumumab + Osimertinib | Cohort A: Ramucirumab + Osimertinib
Started | 3 | 4 | 22
Received at Least One Dose of Study Drug | 3 | 4 | 22
Completed | 0 | 1 | 5
Not Completed | 3 | 3 | 17
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Progressive Disease | 1 | 3 | 14

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Arm B: Necitumumab + Osimertinib: Participants received Necitumumab 800 mg given IV on Days 1 and 8 every 3 weeks and osimertinib 80 mg given orally daily during each 21 day cycle. All participants were treated until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
- Total: Total of all reporting groups
Arm/Group | Arm A: Ramucirumab + Osimertinib | Arm B: Necitumumab + Osimertinib | Cohort A: Ramucirumab + Osimertinib | Total
Number analyzed (Participants) | 3 | 4 | 22 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 12 | 16
  >=65 years | 1 | 2 | 10 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 17 | 21
  Male | 2 | 1 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 22 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 13 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 4 | 9 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 0 | 6 | 6
  United States | 1 | 1 | 3 | 5
  Taiwan | 0 | 0 | 5 | 5
  France | 0 | 1 | 0 | 1
  Spain | 2 | 2 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A Dose Limiting Toxicity (DLT) was defined as one of the following Adverse Events (AE) that is likely related to the study drug or combination, and fulfils any one of the following criteria, graded according to the NCI-CTCAE Version 4.0:
  1. Any nonhematologic Grade ≥3 toxicity, except for toxicities such as liver or renal function abnormality, skin rash that resolves with appropriate therapy, transient hypersensitivity and injection site reactions, myalgia, fatigue, constipation, electrolyte imbalance, nausea, vomiting, diarrhea
  2. Hematologic toxicity was considered a DLT as the following:
     1. Grade 4 toxicity lasting ≥7 days, or
     2. Grade 3 or 4 thrombocytopenia if associated with bleeding or requires platelet transfusion, or
     3. Febrile neutropenia
  3. Death if considered related to study treatment
  4. Any other significant toxicity deemed by the primary investigator and Lilly clinical research personnel to be dose limiting
Time Frame: Arm A: Cycle 1 through Cycle 2 (14-day cycle); Arm B: Cycle 1 (21-day cycle)
Population: Arm A: participants who either completed the first 2 cycles of treatment or discontinued from study treatment or study participation Arm B: participants who either completed the first cycle of treatment or discontinued from study treatment or study participation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ramucirumab + Osimertinib | Arm B: Necitumumab + Osimertinib
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Description: Cmin was the concentration of study drug in the blood immediately before the next dose was administered.
Time Frame: Predose on Day (D) 1 of Cycle (C) 2, Predose on Day 1 of Cycle 4, Predose on Day 1 of Cycle 5, Predose on Day 1 of Cycle 7, Predose on Day 1 of Cycle 13
Population: All enrolled participants who received at least one dose of ramucirumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- Arm A/Cohort A: Ramucirumab + Osimertinib: Participants received Ramucirumab 10 mg/kg given IV on Day 1 every 2 weeks and osimertinib 80 mg given orally daily during each 14-day cycle. All participants were treated until confirmed progressive disease, unacceptable toxicity, or discontinuation for any other reason.
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 20
microgram per milliliter (µg/mL)
  D1C2 | 41.3 (56.3)
  D1C4: number analyzed (Participants) | 16
  D1C4 | 66.7 (34.3)
  D1C5: number analyzed (Participants) | 15
  D1C5 | 76.7 (27)
  D1C7: number analyzed (Participants) | 10
  D1C7 | 90.7 (26.6)
  D1C13: number analyzed (Participants) | 4
  D1C13 | 103 (29.6)

3. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab
Description: Cmin was the concentration of study drug in the blood immediately before the next dose was administered.
Time Frame: Predose on Day 1 of Cycle 3, Predose on Day 1 of Cycle 5
Population: All enrolled participants who received at least one dose of necitumumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Arm B: Necitumumab + Osimertinib
Number analyzed (Participants) | 2
nanograms per milliliter (ng/mL)
  D1C3 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there were only two participants. Individual values reported: 575476.3 ng/mL and 150490.8 ng/mL
  D1C5: number analyzed (Participants) | 1
  D1C5 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 225257.8 ng/mL

4. Secondary Outcome: Objective Response Rate (ORR) for Ramucirumab in Combination With Osimertinib: Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: ORR was the best overall response of complete response (CR) or partial response (PR) as classified by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). CR was a disappearance of all target and non-target lesions and normalization of tumor marker level. PR was an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression (up to 25 months)
Population: All enrolled participants from the ramucirumab + osimertinib arms who received at least one dose of study drug. Per Protocol, the outcomes for a combination of ramucirumab and osimertinib were analyzed under a single arm (Arm A/Cohort A), as Cohort A is an extension of Arm A.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 25
Percentage of Participants | 76 [58.1 to 89.0]

5. Secondary Outcome: Disease Control Rate (DCR) for Ramucirumab in Combination With Osimertinib: Percentage of Participants With CR, PR or Stable Disease (SD)
Description: DCR was the best overall response of CR, PR, or SD as defined by RECIST v1.1. CR was defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or one or more new lesions.
Time Frame: Baseline to Objective Disease Progression (up to 25 months)
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 25
Percentage of Participants | 92 [76.9 to 98.6]

6. Secondary Outcome: Duration of Response (DoR) for Ramucirumab in Combination With Osimertinib
Description: Duration of Response (DoR) was defined only for participants with a confirmed CR or PR. It was measured from the date of first evidence of a confirmed CR or PR to the date of objective progression or the date of death due to any cause, whichever is earlier. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date, DOR was censored at the date of the last complete objective progression-free disease assessment.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death from Any Cause (up to 25 months)
Population: All enrolled participants from the ramucirumab + osimertinib arms who received at least one dose of study drug with a confirmed CR or PR (including censored). Number of participants censored = 7.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 19
Months | 13.37 [9.63 to 21.19]

7. Secondary Outcome: Progression Free Survival (PFS) for Ramucirumab in Combination With Osimertinib
Description: Progression-free survival (PFS) was the time from the date of first study treatment until the date of radiographic documentation of progression (as defined by RECIST v. 1.1) based on investigator assessment or the date of death due to any cause, whichever was earlier. If a participant did not have a complete baseline disease assessment, then the PFS time was censored at the enrollment date, regardless of whether or not objectively determined disease progression or death was observed for the participant; otherwise, if a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last complete objective progression-free disease assessment date.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (up to 26 months)
Population: All enrolled participants from the ramucirumab + osimertinib arms who received at least one dose of study drug (including censored). Number of participants censored = 7.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 25
Months | 11.04 [5.49 to 19.29]

8. Secondary Outcome: Overall Survival (OS) for Ramucirumab in Combination With Osimertinib
Description: OS was date of first study treatment until death due to any cause. If the participant was alive at the data inclusion cutoff date for the analysis (or was lost to follow-up), OS was censored on the last date the participant was known to be alive.
Time Frame: Baseline to Death from Any Cause (up to 29 months)
Population: All enrolled participants from the ramucirumab + osimertinib arms who received at least one dose of study drug (including censored). Number of participants censored = 13.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm A/Cohort A: Ramucirumab + Osimertinib
Number analyzed (Participants) | 25
Months | NA [16.03 to NA] — There were not enough events to estimate the median, upper confidence limit.

ADVERSE EVENTS:
Time Frame: Baseline to follow up (5.38 years)
Description: All enrolled participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Arm A: Ramucirumab + Osimertinib | Arm B: Necitumumab + Osimertinib | Cohort A: Ramucirumab + Osimertinib
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 11/22
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 8/22
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ramucirumab + Osimertinib (N=3) | Arm B: Necitumumab + Osimertinib (N=4) | Cohort A: Ramucirumab + Osimertinib (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A: Ramucirumab + Osimertinib (N=3) | Arm B: Necitumumab + Osimertinib (N=4) | Cohort A: Ramucirumab + Osimertinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Trichomegaly (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (19) | 14 (38)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 8 (11)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (16)
Transient lingual papillitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (9)
Asthenia (General disorders) | 1 (2) | 1 (11) | 2 (3)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 3 (3) | 3 (6)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2) | 3 (5)
Non-cardiac chest pain (General disorders) | 1 (2) | 1 (2) | 3 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 5 (10)
Pain (General disorders) | 0 (0) | 1 (2) | 4 (4)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 3 (3)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 3 (10)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (7)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 4 (13)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 1 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (20)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 6 (49)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 3 (19)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 9 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (6)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 9 (11)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 4 (8)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/17 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 6 (8)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (24)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (6)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (12) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 2 (3)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1/3 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (9)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (9) | 4 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 14 (24)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT02789345/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT02789345/SAP_001.pdf